CLINICAL TRIAL: NCT03809299
Title: 2-A-Day Study: Twice a Day Meals Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-9671; 5P30DK020541 (NIH)
Record Dates: First submitted 2019-01-08; First posted 2019-01-18 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: PreDiabetes
Keywords: Caloric restriction; Fasting; intermittent fasting; isocaloric ad lib meal timing; Twice-a-day feeding; insulin; glucose metabolism; normoglycemia; hyperglycemia
MeSH Terms: conditions — Prediabetic State; Fasting; Intermittent Fasting; Insulin Resistance; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ad libitum meal timing first (Other): This arm will receive the ad libitum meal timing intervention first, followed by the twice a day feeding intervention.
  Interventions: Other: Ad libitum meal timing; Other: Twice a day meals
- Twice a day meals first (Other): This arm will receive the twice a day feeding intervention first, followed by the ad libitum meal timing intervention.
  Interventions: Other: Ad libitum meal timing; Other: Twice a day meals

INTERVENTIONS:
Other: Ad libitum meal timing — Research participants will eat meals provided by the study throughout the day, ad libitum
Other: Twice a day meals — Research participants will eat meals provided by the study at two intervals during the day, and fast in between.

SUMMARY:
Caloric restriction increases lifespan and/or healthspan across multiple species. However implementation of long-term CR in humans is problematic and unacceptable to many individuals. As a result, intermittent fasting models have been developed to improve adherence. Such models have been shown to improve blood pressure, insulin sensitivity, decrease hepatic fat content and body weight. Investigators established an isocaloric twice-a-day (ITAD) feeding plan in mice, wherein test mice were acclimatized to consume over two hour periods (8-10am and 5-7pm), the same amount of food as ad-libitum mice. This intervention prevented obesity and age-associated type 2 diabetes via system-wide activation of autophagy. The investigators will perform further studies of the same feeding model in humans in a randomized crossover design. The objective is to test the hypothesis that restricting eating periods to twice a day (TAD), when compared to isocaloric ad lib meal timing (ALMT), will have beneficial effects on glucose metabolism, body composition, energy expenditure and autophagy in human subjects at risk for diabetes

DETAILED DESCRIPTION:
Caloric restriction (CR) increases lifespan and/or healthspan across multiple species including non-human primates. However, implementation of long-term CR in humans is problematic and unacceptable to many individuals. Further, since CR leads to loss of muscle mass in mice, it is likely that its implementation as a restorative strategy during aging may exacerbate age-associated muscle loss. As a result, intermittent fasting models, e.g., alternate-day fasting, alternate day-modified fasting, the 5:2 diet, and the more recently elucidated early time-restricted feeding (eTRF)3 were developed as alternative strategies to improve adherence. Intermittent fasting increases glucose clearance/improves insulin sensitivity, decreases hepatic fat content, lowers blood pressure and body weight by varying degrees (at least when calories were unmatched). Despite these metabolic advantages, these approaches have also shown poor adherence in humans. For instance, alternate-day fasted subjects remained hungry on the fast days, which led to the conclusion that this approach cannot be continued for extended periods of time, and that adding one small meal on the fasting day may make this model more acceptable. Accordingly, in alternate day-modified fasting, fasted days (25% caloric intake) alternated with feasting days (125% calories), which improved compliance although dropout rates remained relatively high (38%) when compared to control group (26%). In addition, this feeding approach was not found to be superior to daily caloric restricted controls in terms of adherence, weight loss or cardiovascular benefits. More recently, eTRF wherein men with prediabetes were subjected to a 6-hr feeding interval with dinner before 1 pm displayed a number of metabolic benefits when compared to individuals on a 12-hr feeding time-frame. Nevertheless, due to vocational or societal factors, it is plausible that a vast majority of individuals may not be able to adhere to a regimen requiring the consumption of three meals within the first 6 hr of the diurnal cycle. In the attempt to offset compliance-related issues and to pursue a simpler approach, investigators established an isocaloric twice-a-day (ITAD) feeding plan in mice, wherein test mice are acclimatized to consume over two 2hr-periods (8:00-10:00am and 5:00-7:00pm) the same amount of food as ad libitum-fed mice. This would effectively translate to a breakfast and dinner (two meals) in humans. It has been shown that two periods of food restriction per day in mice prevents obesity and age-associated type 2 diabetes via system-wide activation of autophagy. This study is to determine if twice-a-day feeding will restore normoglycemia and promote metabolic correction in older men with prediabetes.

Autophagy is a lysosomal degradative pathway that plays key roles in maintaining "clean" cells. It is well-established that basal autophagy levels begin to decline progressively in aged organisms. Maintaining higher autophagy levels improves organ function and stress response. For instance, liver-specific overexpression of autophagy genes protects against diet-induced obesity and tumor necrosis factor-mediated acute hepatotoxicity. In the investigators' studies with ITAD feeding in mice, blocking autophagy in distinct tissues resulted in loss of the metabolic benefits from this feeding strategy. Consequently, it is propose that establishing ITAD feeding in humans will yield a cost-effective, practical and immediately translatable strategy to prolong health-span by preventing diabetes and sarcopenia as well as the vast number of secondary diseases caused by sustained hyperglycemia.

This study will investigate the feasibility of a TAD eating regimen and collect preliminary data to inform a larger-scale and more definitive trial.

Specific Aims:

Aim 1: To assess the feasibility of implementing a structured TAD eating regimen using study-provided meals 1a. To design meal plans that are isocaloric with habitual intake and intended to maintain weight and to develop methods to prepare, package and deliver the meals.

1b. To develop and evaluate methods to enhance and monitor participant adherence to TAD eating; this will include patient logs, photo records of food intake and continuous (participant blinded) glucose monitoring.

1. c. To assess participant satisfaction with TAD meal restriction, using validated instruments to evaluate hunger, satiety and well-being Aim 2: To collect preliminary data on the effect of TAD meal restriction to inform design of an adequately powered RCT
2. a. To collect preliminary data on the effect of TAD meal restriction on glucose tolerance, insulin sensitivity and secretion, body composition and energy expenditure

2b. To collect preliminary data on the effect of TAD meal restriction on cellular processes related to autophagy

ELIGIBILITY:
Inclusion Criteria:

* ● Men, age 30-70 years. In this preliminary study, recruitment is limited to men because data from the relevant animal studies showed marked sexual dimorphism, with more pronounced metabolic effects in males. Future studies will include both males and females.

  * IFG or IGT based on 75g OGTT (fasting plasma glucose 100 -125 mg/dl and/or 2-hr glucose between 140 - 199 mg/dl); Or diabetes (FPG > 126 mg/dl or 2 hr glucose > 200 mg/dl) not on treatment and with HbA1c < 6.8% can also be enrolled.

    * BMI 25-35 kg/m2

Exclusion Criteria:

* Type 2 diabetes with A1C ≥6.8% or on drug treatment; Type 1 diabetes
* Treatment with drugs known to influence glucose metabolism (diabetes medications, systemic glucocorticoids, niacin > 500 mg/day)
* Current smoking, alcohol or drug abuse
* Vigorous habitual physical activity (e.g., marathon runner, heavy weights trainers)
* Subjects with symptomatic gastrointestinal disorders or intolerance (e.g., food allergies, lactose intolerance, gluten sensitivity, etc.) or other conditions requiring special diet or meal timing.
* Subjects with serious chronic illness: severe (activity limiting) COPD, NYHA class 3 or 4 heart failure, kidney disease (eGFR<45ml/min), liver enzyme abnormalities (ALT > 2 times ULN), stroke, MI or ACS within last 6 months, cancer or HIV disease under treatment.
* Any other disease/condition that the investigator believes may interfere with participation in the study (e.g., eating disorder).
* Unstable weight conditions: gain or loss of > 5 pounds or 2.5% body weight in past 3 months.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 5 weeks
  insulin sensitivity as measured by the Matsuda Index

SECONDARY OUTCOMES:
Glucose tolerance | 5 weeks
  Glucose level after oral glucose tolerance test as measured by glucose area under the curve.
Body Composition | 5 weeks
  Fat mass as estimated by bioimpedance analysis
Energy expenditure | 5 weeks
  Resting energy expenditure as estimated by indirect calorimetry
Autophagy level | 1 week
  Expression of levels of autophagosome marker LC3 by immunoblotting

CONTACTS AND LOCATIONS:
Overall Officials: Jill Crandall, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No